CLINICAL TRIAL: NCT04543019
Title: Age, Body Mass Index and Tumor Sidedness in Metastatic Colorectal Cancer Patients as Predictive Factors for Systemic Therapy Outcome
Brief Title: Effect of Age, Body Mass Index and Tumor Sidedness in Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehad Ahmed Abd El-Razik, principal investigator, Assiut University
Other Study IDs: systemic therapy in mCRC
Record Dates: First submitted 2020-08-20; First posted 2020-09-09 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine progression free survival (PFS) and overall survival (OS) in metastatic colorectal cancer in relation to age, BMI and tumor sidedness, describing their predictive influence on systemic therapy outcome.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) represents a major public health concern as it is the third most frequently diagnosed cancer and the fourth cause of cancer-related mortality worldwide . The ﬁve-year survival rate is around 64.9% for all stages, while in metastatic cases, it only reaches 13.1% .

Approximately 26% of CRCs are diagnosed at stage IV among patients aged younger than 50 years, compared with 23% in those aged 50 to 64 years and 19% among those aged 65 years and older. Overall survival (OS) among patients younger than 50 years (68%) is similar to that in those 50 to 64 years (69%) because of a later stage at diagnosis.

Obesity is associated with an increased incidence of CRC . In recent studies body mass index (BMI) was prognostic for overall survival and progression free survival. That is risk of progression and/or death was greatest for low BMI; risk decreased as BMI increased. BMI was not predictive of treatment effect . Cachexia and associated poor performance status have previously been identiﬁed as negative prognostic factors in patients with CRC.

Tumor sidedness is an independent prognostic factor in patients with early and metastatic CRC as left-sided primaries have improved outcomes. sidedness also represents a powerful predictor of benefit from anti epidermal growth factor receptor[EGFR] inhibitors therapies in patients with RAS wild-type metastatic CRC (mCRC) .

The mainstay of treatment of mCRC includes cytotoxic chemotherapy with the addition of a molecularly targeted agent . The cytotoxic regimens that are usually used include a combination of oxaliplatin or irinotecan with a fluoropyrimidine, in addition to targeted agents such as [EGFR] inhibitors for patients with RAS wild-type mCRC or vascular endothelial growth factor inhibitors .

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Pathologically proven colon or rectal adenocarcinoma.
* Stage IV colorectal cancer.

Exclusion Criteria:

* Age <18 years.
* Not pathologically proven colon or rectal adenocarcinoma.
* Stage I, II and III colorectal cancer.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Total coverage sample will be used. Fifty patients having the inclusion criteria who presented to Clinical oncology department, Assiut university hospital between January 2015 to December 2019 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) and overall survival (OS) | between January 2015 and December 2019
  Progression free survival (PFS) and overall survival (OS) in metastatic colorectal cancer patients in correlation to age, BMI and tumor sidedness.

SECONDARY OUTCOMES:
response to systemic therapy | between January 2015 and December 2019
  response to systemic therapy in correlation to age, BMI and tumor sidedness

REFERENCES:
- [Background] Yoshino T, Arnold D, Taniguchi H, Pentheroudakis G, Yamazaki K, Xu RH, Kim TW, Ismail F, Tan IB, Yeh KH, Grothey A, Zhang S, Ahn JB, Mastura MY, Chong D, Chen LT, Kopetz S, Eguchi-Nakajima T, Ebi H, Ohtsu A, Cervantes A, Muro K, Tabernero J, Minami H, Ciardiello F, Douillard JY. Pan-Asian adapted ESMO consensus guidelines for the management of patients with metastatic colorectal cancer: a JSMO-ESMO initiative endorsed by CSCO, KACO, MOS, SSO and TOS. Ann Oncol. 2018 Jan 1;29(1):44-70. doi: 10.1093/annonc/mdx738. PMID 29155929
- [Background] El-Deiry WS, Vijayvergia N, Xiu J, Scicchitano A, Lim B, Yee NS, Harvey HA, Gatalica Z, Reddy S. Molecular profiling of 6,892 colorectal cancer samples suggests different possible treatment options specific to metastatic sites. Cancer Biol Ther. 2015;16(12):1726-37. doi: 10.1080/15384047.2015.1113356. PMID 26553611
- [Background] Labianca R, Nordlinger B, Beretta GD, Mosconi S, Mandala M, Cervantes A, Arnold D; ESMO Guidelines Working Group. Early colon cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi64-72. doi: 10.1093/annonc/mdt354. No abstract available. PMID 24078664
- [Background] Murphy CC, Harlan LC, Lund JL, Lynch CF, Geiger AM. Patterns of Colorectal Cancer Care in the United States: 1990-2010. J Natl Cancer Inst. 2015 Jul 23;107(10):djv198. doi: 10.1093/jnci/djv198. Print 2015 Oct. PMID 26206950
- [Background] Larsson SC, Wolk A. Obesity and colon and rectal cancer risk: a meta-analysis of prospective studies. Am J Clin Nutr. 2007 Sep;86(3):556-65. doi: 10.1093/ajcn/86.3.556. PMID 17823417
- [Background] Renfro LA, Loupakis F, Adams RA, Seymour MT, Heinemann V, Schmoll HJ, Douillard JY, Hurwitz H, Fuchs CS, Diaz-Rubio E, Porschen R, Tournigand C, Chibaudel B, Falcone A, Tebbutt NC, Punt CJ, Hecht JR, Bokemeyer C, Van Cutsem E, Goldberg RM, Saltz LB, de Gramont A, Sargent DJ, Lenz HJ. Body Mass Index Is Prognostic in Metastatic Colorectal Cancer: Pooled Analysis of Patients From First-Line Clinical Trials in the ARCAD Database. J Clin Oncol. 2016 Jan 10;34(2):144-50. doi: 10.1200/JCO.2015.61.6441. Epub 2015 Oct 26. PMID 26503203
- [Background] Argiles JM, Busquets S, Stemmler B, Lopez-Soriano FJ. Cancer cachexia: understanding the molecular basis. Nat Rev Cancer. 2014 Nov;14(11):754-62. doi: 10.1038/nrc3829. Epub 2014 Oct 9. PMID 25291291
- [Background] Tisdale MJ. Cachexia in cancer patients. Nat Rev Cancer. 2002 Nov;2(11):862-71. doi: 10.1038/nrc927. No abstract available. PMID 12415256
- [Background] Thoresen L, Frykholm G, Lydersen S, Ulveland H, Baracos V, Prado CM, Birdsell L, Falkmer U. Nutritional status, cachexia and survival in patients with advanced colorectal carcinoma. Different assessment criteria for nutritional status provide unequal results. Clin Nutr. 2013 Feb;32(1):65-72. doi: 10.1016/j.clnu.2012.05.009. Epub 2012 Jun 12. PMID 22695408
- [Background] Petrelli F, Tomasello G, Borgonovo K, Ghidini M, Turati L, Dallera P, Passalacqua R, Sgroi G, Barni S. Prognostic Survival Associated With Left-Sided vs Right-Sided Colon Cancer: A Systematic Review and Meta-analysis. JAMA Oncol. 2017 Feb 1;3(2):211-219. doi: 10.1001/jamaoncol.2016.4227. PMID 27787550
- [Background] Van Cutsem E, Oliveira J; ESMO Guidelines Working Group. Advanced colorectal cancer: ESMO clinical recommendations for diagnosis, treatment and follow-up. Ann Oncol. 2009 May;20 Suppl 4:61-3. doi: 10.1093/annonc/mdp130. No abstract available. PMID 19454465
- [Background] Hochster HS, Grothey A, Hart L, Rowland K, Ansari R, Alberts S, Chowhan N, Ramanathan RK, Keaton M, Hainsworth JD, Childs BH. Improved time to treatment failure with an intermittent oxaliplatin strategy: results of CONcePT. Ann Oncol. 2014 Jun;25(6):1172-8. doi: 10.1093/annonc/mdu107. Epub 2014 Mar 7. PMID 24608198